CLINICAL TRIAL: NCT05210855
Title: Comparison of Image Quality Between Ultra-low Dose (ULD) and Standard Dose CT Scans in Detecting Traumatic Brain Injury in the Emergency Room
Acronym: ULD-CRANE 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NIMAO/2020-1/NM-02
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Closed Head Injury; Penetrating Head Injury
MeSH Terms: conditions — Head Injuries, Closed; Head Injuries, Penetrating | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with head trauma (Experimental)
  Interventions: Diagnostic Test: CT scan

INTERVENTIONS:
Diagnostic Test: CT scan — Scan with classic dose followed by ultra-low dose

SUMMARY:
Head trauma is a frequent reason for consultation in the emergency room. The CT scan is the reference examination allowing rapid management of the patient. However, CT examinations are among the diagnostic examinations with the highest exposure to ionizing radiation. The study investigators have previously implemented "ultra-low dose" (ULD) acquisitions for several pathologies with an effective dose level similar to that of a standard radiographic examination. These ULD acquisitions are now routinely used in our clinical practice for explorations of the thorax, spine, pelvis and proximal femurs, extremities.

This study expands these ULD acquisitions to skull CT for detecting traumatic intracranial lesions.

The study investigators hypothesize that it would be possible to search for intracranial lesions in patients with head trauma using ULD protocols, thereby reducing the doses delivered to the patient while maintaining sufficient image quality for the diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting to the emergency room of the CHU of Nîmes for a cranial trauma requiring scanning.
* Patient with isolated head injury or polytrauma patient with head injury among others.
* The patient or their legal representative or family member must have given their free and informed consent and signed the consent form, or the patient was included under an emergency situation
* The patient must be a member or beneficiary of a health insurance plan

Exclusion Criteria:

* The subject is participating in a study prohibiting participation in other studies, or is in a period of exclusion determined by a previous study
* Patient is pregnant, parturient or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

PRIMARY OUTCOMES:
Image quality of ultra-low dose scan compared to classic dose for visualising the differentiation of grey/white matter | Day 0
  5-point scale: unacceptable, sub-optimal, acceptable, better than average
Image quality of ultra-low dose scan compared to classic dose for visualising lenticular nuclei | Day 0
  5-point scale: unacceptable, sub-optimal, acceptable, better than average
Image quality of ultra-low dose scan compared to classic dose for visualising the ventricular system | Day 0
  5-point scale: unacceptable, sub-optimal, acceptable, better than average
Image quality of ultra-low dose scan compared to classic dose for visualising basal cisterns | Day 0
  5-point scale: unacceptable, sub-optimal, acceptable, better than average
Image quality of ultra-low dose scan compared to classic dose for visualising deconvexed subarachnoid spaces | Day 0
  5-point scale: unacceptable, sub-optimal, acceptable, better than average

SECONDARY OUTCOMES:
Inter-evaluator concordance (senior versus junior) in visualizing all five structures (differentiation of grey/white matter, lenticular nuclei, ventricular system, basal cisterns, deconvexed subarachnoid spaces) | Day 0
  Total score of the 5 Likert scores
Presence of at least one extradural hematoma by ultra-low dose versus classical scanner | Day 0
  Yes/no
Presence of at least one subarachnoid hemorrhage by ultra-low dose versus classical scanner | Day 0
  Yes/no
Presence of at least one subdural hematoma by ultra-low dose versus classical scanner | Day 0
  Yes/no
Presence of at least one intraparenchymal hemorrhage by ultra-low dose versus classical scanner | Day 0
  Yes/no
Presence of at least one intracranial hemorrhage by ultra-low dose versus classical scanner | Day 0
  Yes/no
Presence of at least one cranial bone lesion by ultra-low dose versus classical scanner | Day 0
  Yes/no
Presence of at least one bone lesion by ultra-low dose versus classical scanner | Day 0
  Yes/no
Radiologist-reported image quality of ultra-low dose versus classical scanner | Day 0
  4-point Likert scale: Interpretable, interpretable despite moderate technical issues (centering, movement, constant), entirely interpretable despite moderate technical issues (centering, movement, constant), No technical issues
Radiologist-reported diagnostic quality of ultra-low dose versus classical scanner | Day 0
  4-point Likert scale: unacceptable, sub-optimal, acceptable, better than average
Radiologist-reported confidence level of ultra-low dose versus classical scanner | Day 0
  4-point Likert scale: unacceptable, sub-optimal, acceptable, better than average
Interpretation time of ultra-low dose versus classical scanner for a senior and junior evaluator | Day 0
  Minutes

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Menjot de Champfleur, Principal Investigator — CHU Nimes
Locations (1):
- CHU de Nimes, Nîmes, France